CLINICAL TRIAL: NCT00620737
Title: Pilot Safety and Efficacy Study of Isolagen Therapy in Treatment of Restrictive Burn Scars
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company Decision
Sponsor: Castle Creek Biosciences, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IT-B-001
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Restrictive Burn Scars of Joint Area

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Arm (Experimental): Active Treatment
  Interventions: Biological: Autologous Human Fibroblasts (Isolagen TherapyTM)
- Control Arm (Placebo Comparator): Placebo treatment
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Autologous Human Fibroblasts (Isolagen TherapyTM) — 1. Collection of skin biopsy.
  2. Administration of 2 study injections
  3. Performance of various study assessments during clinic visits
  Arms: Active Arm
Biological: Placebo — 1. Collection of skin biopsy.
  2. Administration of 2 study injections
  3. Performance of various study assessments during clinic visits
  Arms: Control Arm

SUMMARY:
The purpose of this study is to evaluate the safety profile and the treatment effect of Isolagen TherapyTM and placebo when administered to stable restrictive burn scars of an affected joint area.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age
* Subject has "stable" restrictive burn scar of a jointed area that restricts range of motion (ROM) of the affected joint by greater than or equal to 20% and that is no deeper than the fascia (i.e., underlying structures including ligament, tendon, muscle, and bone must not contribute to the restriction)
* Subject agrees to maintain any current physical therapy regimen for the duration of the study
* Subject must be able to provide written informed consent and comply with the study requirements
* Females of childbearing potential must have a negative urine pregnancy test at the screening visit and must agree to use a reliable means of birth control for the duration of the study
* Male subjects must agree to use a reliable means of birth control for the duration of the study
* Subject has healthy, non-scarred post auricular, abdomen, back of neck at hairline, lower abdomen, upper arm, side of upper leg, or axillary region (on the lateral thorax) skin area suitable for biopsy
* Subject has normal CBC, thyroid function, renal function, liver function, blood glucose and SMA 18 at Screening

Exclusion Criteria:

* The restrictive burn scar to be treated is primarily classified as a keloid scar
* Surgical release of scar to be treated within the last 12 months
* Subjects for whom a skin biopsy cannot be collected
* Plans to initiate any new scar therapy during the study period
* Treatment with an investigational product or procedure within 30 days prior to study enrollment or plans to participate in another clinical trial during the course of this study
* History of active autoimmune disease or organ transplantation
* Diagnosis of cancer, including basal cell carcinoma, unless successfully treated or in remission for a minimum of 6 months
* Known genetic disorders affecting fibroblasts or collagen, such as achondroplasia, osteogenesis imperfecta, epidermolysis bullosa, ataxia-telangiectasia, or Ehlers Danlos syndrome
* Active systemic infection as shown by any one of the following: symptoms, fever and/or an elevated white count (subjects who present with an active systemic infection may be enrolled and biopsied after the infection has resolved)
* Requires chronic antibiotic or steroidal therapy
* Any conditions that are considered by the Investigator to be contraindications to biopsy or injection
* Pregnant or lactating women or women trying to become pregnant during the study
* Subject has any disorder that may prevent compliance, such as history of chronic alcohol or drug abuse, significant mental or nervous disorder or other illness that would, in the Investigator's opinion, interfere with the study
* Presence of other disease or condition that would result in impairment of the range of motion of the extremity, e.g. rheumatoid arthritis or stroke
* Subjects with a known allergy to gentamycin or amphotericin B, or sensitivity to materials of bovine origin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of all study assessments | Day 0, 14, 30, 60, 90 and 120

SECONDARY OUTCOMES:
Review of adverse Events, vital signs and physical examination | Day 0, 14, 30, 60, 90 and 120

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Nassau County Medical Center, East Meadow, New York
  - University of Texas Medical Branch- Galveston, Galveston, Texas